CLINICAL TRIAL: NCT01013987
Title: A Phase 4, Single Arm, Open Label, Pilot Study of Maraviroc (Celsentri) in Combination With Raltegravir and Darunavir/Ritonavir for the Treatment of Triple Class Failure in Adult HIV-1 Infected Patients.
Brief Title: Maraviroc (Celsentri) With Raltegravir and Darunavir/Ritonavir for the Treatment of Triple Class Failure in Adult HIV-1 Infected Patients
Acronym: TERCETO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Huésped (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Pedro Cahn, Fundación Huésped
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TERCETO
Record Dates: First submitted 2009-11-13; First posted 2009-11-16 (Estimated); Last update posted 2010-02-10 (Estimated); Status verified 2009-11

CONDITIONS: HIV-1 Adults Patients; AIDS; Triple Class Failure
Keywords: HIV-1; triple class failure; Maraviroc; Raltegravir; Darunavir/ritonavir; Maraviroc with raltegravir and darunavir/ritonavir
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Maraviroc; Raltegravir Potassium; Darunavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: maraviroc — maraviroc: one 150 mg pill twice daily
  Other Names: Celsentri
Drug: Raltegravir — raltegravir : one 400 mg pill twice daily
  Other Names: Issentres
Drug: Darunavir/ritonavir — * darunavir : two 300 mg pills twice daily with meal
  * ritonavir: one 100 mg pill twice daily with meal

SUMMARY:
Phase 4, single arm, open label study designed to compare the safety and efficacy of antiviral activity and immunological effect of Maraviroc in combination with Raltegravir and Darunavir/Ritonavir for treatment of triple class failure in adult HIV-1 infected subjects.

The purpose of this study is to look at the safety and efficacy of a combination of 3 new antiretroviral drugs: maraviroc, darunavir and raltegravir in patients who have multi-resistant viruses and limited treatment options. Patients will undergo treatment for 48 weeks; safety and virological efficacy will be preliminary evaluated at weeks 16 and 24.

DETAILED DESCRIPTION:
This is a Phase 4, single arm, open-label, study designed to demonstrate the safety, tolerability, efficacy, antiviral and immunological activity of Maraviroc in combination with Raltegravir and Darunavir/Ritonavir in patients with limited to no treatment option in HIV-1 infected subjects ≥ 21 years old.

The trial population will comprise 60 HIV-infected subjects with history of triple class antiretroviral failure, naïve to CCR5-inhibitors, integrase-inhibitors and darunavir will be evaluated. Single arm, stratified according to plasma viral load at screening (> or < 100,000 copies/ml).

Those with evidence of R5 viruses and susceptibility to darunavir in the resistance testing analysis, plus history of failure to NRTIs, NNRTIs and at least one PI, plus a genotype analysis showing evidence of resistance to NRTIs (at least 2 TAMS and/or Q151M and or 69ss), resistance to PIs (at least 2 major mutations), will start a regimen of maraviroc, raltegravir and ritonavir boosted darunavir.

This trial will consist of a screening period of up to 6 weeks, a 48-week treatment period, with interim analysis at 16 and 24 weeks. Followed by a 4-week post-treatment follow-up (FU) period.

Virologic response, CD4 count change, clinical outcomes and safety will be followed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject is at least 21 years of age.
2. Patient with documented HIV-1 infection defined as a positive ELISA plus a confirmatory Western Blot; or alternatively, a plasma HIV- RNA ≥10,000 copies/ml ever documented.
3. Subject has voluntarily signed and dated an informed consent form, approved by an Institutional Review Board (IRB)/Independent Ethics Committee (IEC), after the nature of the study has been explained and the subject has had the opportunity to ask questions. The informed consent must be signed before any study-specific procedures are performed.
4. Subject agrees not to take any medication during the study, including over the counter medicines, vitamins, minerals, herbal preparations, alcohol or recreational drugs without the approval of the trial physician.
5. Documented HIV RNA >500 copies/ml
6. Subject triple class antiretroviral failure (NRTI, NNRTI, PI)
7. Subject naïve to CCR5-inhibitors, integrase-inhibitors and darunavir.
8. Subjects can comply with protocol requirements.
9. Subject's general medical condition, in the investigator's opinion, does not interfere with assessments and completion of the trial.
10. If female, subject must be either postmenopausal for at least one year, surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy), or she must:

    1. use of a double birth control method that includes at least one barrier method, that is acceptable to both the subject and investigator, and
    2. has a urine pregnancy test performed at the Screening Visit and on Baseline, and results of both tests must be negative.
    3. continue practicing birth control methods for at least 30 days after the end of the treatment period.
11. Subject present R5 HIV1 at Screening, verified by Trofile Essay by Monogram Bioscience.

Exclusion Criteria:

1. Evidence of resistance against Maraviroc, Raltegravir, Darunavir/Ritonavir, based on the resistance test performed at Screening.
2. Previously documented HIV-2 infection.
3. Use of disallowed concomitant therapy listed in guidelines for use of each drug.
4. Patient has a current (active) diagnosis of acute hepatitis due to any cause OR chronic hepatitis B and/or C WITH aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT)>5 x upper limit of normal (ULN) AND/OR is likely to require treatment in the next year.
5. Any active clinically significant disease (e.g. tuberculosis, cardiac disfunction, pancreatitis) or findings during screening of medical history or physical examination that, in the investigator´s opinion, would compromise the subject´s safety or outcome of the trial or adherence to the trial protocol.
6. Subject has a currently active AIDS defining illness (Category C conditions according to the CDC Classification System for HIV infection 1993) within 30 days of screening. Subjects who are on stable maintenance therapy for an opportunistic infection may be enrolled.
7. Life expectancy < 1 year according to the judgment of the investigator.
8. Screening laboratory analysis show any of the following abnormal laboratory results:

   1. Hemoglobin < 8.0 g/dL
   2. Absolute neutrophil count < 750 cells/µL
   3. Platelet count < 50,000 mm3
9. Subject enrolled in other clinical trials that include any blood sampling, specimen collection, or other interventional procedure. Concurrent participation in non-interventional observational trials
10. Use of any investigational agents within 30 days prior to screening.
11. Use of immunosuppressive drugs, cytokine inhibitors or other cytokines in the last year.
12. Any condition (including but not limited to alcohol and drug use) which in the opinion of the investigator, could compromise the subject's safety or adherence to the protocol;.
13. Subject is pregnant or breast-feeding

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-02

PRIMARY OUTCOMES:
Proportion of patients with HIV RNA levels of less than 50 copies/ml in an intent to treat analysis at week 24 | week 24

SECONDARY OUTCOMES:
Proportion of patients with HIV RNA levels of less than 50 copies/ml at week 24 and with HIV RNA levels of less than 400 copies/ ml at weeks 24 and 48. | week 24 and week 48

CONTACTS AND LOCATIONS:
Locations (1):
- Fundación Huésped, Ciudad de Buenos Aires, Argentina